CLINICAL TRIAL: NCT05565924
Title: Effect of Antigravity Treadmill Training on the Gait Performance and Functional Balance in Patients With Diabetic Peripheral Neuropathy. Randomized Controlled Trial
Brief Title: Alter-G Training on Gait and Balance in Diabetic Neuropathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Ashraf Abdelaal, Associate Professor, Umm Al-Qura University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 13-MED1319-10_IR1
Record Dates: First submitted 2022-06-10; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetic neuropathy; Gait; Balance
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Weight-Bearing; Drug Therapy; Biguanides; Sulfonylurea Compounds; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group-A (Experimental): This group received moderate-intensity (50-70% heart rate reserve) aerobic exercise training on the antigravity treadmill (100% weight-bearing; n=14) 3 times/week for 12-weeks, plus oral drug therapy (Biguanide alone or "Sulfonylureas plus Biguanide combination").
  Interventions: Other: Group- A (100% weight-bearing; n=14), (moderate-intensity (50-70% heart rate reserve) aerobic exercise training on the antigravity treadmill, 3 times/week for 12-weeks.
- Group-B (Experimental): This group received moderate-intensity (50-70% heart rate reserve) aerobic exercise training (70% weight-bearing; n=13) on the antigravity treadmill (AlterG Pro 200, AlterG Inc, California, USA) 3 times/week for 12 weeks, plus oral drug therapy (Biguanide alone or "Sulfonylureas plus Biguanide combination").
  Interventions: Other: Group- B (70% weight-bearing), (moderate-intensity (50-70% heart rate reserve) aerobic exercise training on the antigravity treadmill, 3 times/week for 12-weeks.
- Group-C (Experimental): This group received moderate-intensity (50-70% heart rate reserve) aerobic exercise training (50% weight-bearing; n=14) on the antigravity treadmill (AlterG Pro 200, AlterG Inc, California, USA), 3 times/week for 12 weeks plus oral drug therapy (Biguanide alone or "Sulfonylureas plus Biguanide combination").
  Interventions: Other: Group- C (50% weight-bearing), (moderate-intensity (50-70% heart rate reserve) aerobic exercise training on the antigravity treadmill, 3 times/week for 12-weeks.
- group-D (30% weight-bearing; n=13) (Experimental): This group received moderate-intensity aerobic exercise training (30% weight-bearing; n=13) on the antigravity treadmill (AlterG Pro 200, AlterG Inc, California, USA) 3 times/week for 12 weeks, plus oral drug therapy (Biguanide alone or "Sulfonylureas plus Biguanide combination").
  Interventions: Other: Group- D (30% weight-bearing), (moderate-intensity (50-70% heart rate reserve) aerobic exercise training on the antigravity treadmill, 3 times/week for 12-weeks.
- group-E (control group; n=14) (Sham Comparator): Served as a control group and participated in no aerobic exercise training on the antigravity treadmill (AlterG Pro 200, AlterG Inc, California, USA) during the study, but received oral drug therapy (Biguanide alone or "Sulfonylureas plus Biguanide combination").
  Interventions: Other: Group- E; Control group

INTERVENTIONS:
Other: Group- A (100% weight-bearing; n=14), (moderate-intensity (50-70% heart rate reserve) aerobic exercise training on the antigravity treadmill, 3 times/week for 12-weeks. — Moderate-intensity aerobic exercise training on the antigravity treadmill (100% weight-bearing) plus medications (Biguanide alone or "Sulfonylureas plus Biguanide combination).
  Other Names: Oral drug therapy (Biguanide alone or "Sulfonylureas plus Biguanide combination").
  Arms: Group-A
Other: Group- B (70% weight-bearing), (moderate-intensity (50-70% heart rate reserve) aerobic exercise training on the antigravity treadmill, 3 times/week for 12-weeks. — Moderate-intensity aerobic exercise training on the antigravity treadmill (70% weight-bearing) plus medications plus medications (Biguanide alone or "Sulfonylureas plus Biguanide combination)
  Other Names: Oral drug therapy (Biguanide alone or "Sulfonylureas plus Biguanide combination").
  Arms: Group-B
Other: Group- C (50% weight-bearing), (moderate-intensity (50-70% heart rate reserve) aerobic exercise training on the antigravity treadmill, 3 times/week for 12-weeks. — Moderate-intensity aerobic exercise training on the antigravity treadmill (50% weight-bearing) plus medications (Biguanide alone or "Sulfonylureas plus Biguanide combination)
  Other Names: Oral drug therapy (Biguanide alone or "Sulfonylureas plus Biguanide combination").
  Arms: Group-C
Other: Group- D (30% weight-bearing), (moderate-intensity (50-70% heart rate reserve) aerobic exercise training on the antigravity treadmill, 3 times/week for 12-weeks. — Moderate-intensity aerobic exercise training on the antigravity treadmill (30% weight-bearing) plus medications (Biguanide alone or "Sulfonylureas plus Biguanide combination).
  Other Names: Oral drug therapy (Biguanide alone or "Sulfonylureas plus Biguanide combination").
  Arms: group-D (30% weight-bearing; n=13)
Other: Group- E; Control group — Control: No aerobic exercise training on the antigravity treadmill, but only medications (Biguanide alone or "Sulfonylureas plus Biguanide combination) throughout the study.
  Other Names: Oral drug therapy (Biguanide alone or "Sulfonylureas plus Biguanide combination").
  Arms: group-E (control group; n=14)

SUMMARY:
Diabetic Peripheral Neuropathy and associated complications became globally serious arousing health problems.

Aim: To evaluate the effect of Antigravity treadmill training on gait performance and functional balance in patients with Diabetic Peripheral Neuropathy.

Design: Single-blinded randomized controlled trial. Setting: Outpatient rehabilitation unit. Population: Sixty-eight eligible participants with Diabetic Peripheral Neuropathy were randomly allocated to Five groups: group-A (100% weight-bearing; n=14), group-B (70% weight-bearing; n=13), group-C (50% weight-bearing; n=14), group-D (30% weight-bearing; n=13), group-E (control group; n=14).

Methods: Participants in study groups A, B, C, and D received moderate intensity (50-70% heart rate reserve) aerobic exercise training program on the antigravity treadmill (AlterG, Inc., Fremont, CA, USA) 3 times/week for 12-weeks. The gait performance (using the dynamic gait index) and the functional balance (using the Berg balance scale) variables were evaluated at 3-time points: baseline (evaluation-1), after 12 training weeks (evaluation-2), and 3 months post-training cessation (evaluation-3).

DETAILED DESCRIPTION:
Diabetic Peripheral neuropathy is the most common serious diabetes-related complication affecting more than one-third of patients with diabetes especially those with type 2 diabetes. Diabetic Peripheral neuropathy is defined as the existence of clinical indicators of neural dysfunction after excluding other causes in patients with diabetes and is usually affecting the sensory nerves before the motor ones, following the distal to proximal pattern distribution. Type 2 diabetes-related microangiopathy, neural ischemia, and demyelination are the commonly encountered pathophysiological endpoints responsible for Diabetic Peripheral neuropathy-related neural lesions. The Diabetic Peripheral neuropathy-related proprioceptive inputs impairments further predispose patients to frequently disturbed static and dynamic balance as well as impaired gait performance. Controversy existed regarding the efficacy of the weight-support aerobic exercise training on the locomotion, gait, and functional variables in patients with Diabetic Peripheral neuropathy. Researchers initially thought that weight-bearing exercise training is more beneficial in improving physical function than non-weight-bearing exercise training in patients with Diabetic Peripheral neuropathy. Few studies reported non-significant functional effects of the increased weight support, while others reported beneficial effects of the partial weight off-loading aerobic exercise training on the gait, balance, and functional performance in patients with Diabetic Peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Elderly with diabetic polyneuropathy.
* Diagnosed as having uncontrolled Type 2 Diabetes Mellitus, with glycosylated hemoglobin (HbA1c) levels between 7 and 11 and fasting glucose levels ranging from 7.0 -11.1 mmol/L.
* Treated only with oral anti-diabetic agents (not taking insulin), Pharmacological treatment had to be stable for at least 3 months before the study.
* Able to walk independently with or without an assistive device.
* Scored 19 points or less in the "dynamic gait index.

Exclusion Criteria:

* Type 1 Diabetes Mellitus,
* Patient with malnutrition (Body mass index < 21 kg/m2 or with recent weight loss > 5% body weight in the last month or > 10% in six months).
* Patients With any severe chronic or uncontrolled comorbid condition such as recent myocardial infarction, unstable angina, acute congestive heart failure, third-degree heart block, and uncontrolled arrhythmia.
* Patients will be excluded also if they have abnormal skin integrity e.g. wounds or scar tissues or are on other complementary treatments.
* History of serious cerebrovascular or cardiovascular diseases, and severe debilitating musculoskeletal problems).

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
The gait performance | 12-weeks
  The gait performance (evaluated using the dynamic gait index). The dynamic gait index is composed of eight items/ tasks. According to the participant's performance; each item is scored on a 4-points ordinal scale from 0 to 3; with "0" indicating the worst achievement (severe impairment) while "3" represents the best score (normal performance).
The functional balance | 12-weeks
  The functional balance (evaluated using the Berg balance scale). the Berg balance scale constitutes 14 functional tasks, with each task score ranging from "0 to 4" where "0" indicates the lowest level of function; while "4" indicates the independent performance of the task.

SECONDARY OUTCOMES:
Fasting blood glucose level | 12-weeks
  Fasting blood glucose level

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Abdelaal, Principal Investigator — Umm Al-Qura University
Locations (1):
- Umm Al-Qura University, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No